CLINICAL TRIAL: NCT03349320
Title: Clinical Response to Donepezil in Mild and Moderate Dementia: Relationship to the Drug Plasma Concentration and the CYP2D6 and APOE Genetic Polymorphisms
Brief Title: Response to Donepezil, Drug Plasma Concentration and the CYP2D6 and APOE Genetic Polymorphisms
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Luís Felipe José Ravic de Miranda, Physician, Geriatrician, MD, PhD, Federal University of Minas Gerais
Other Study IDs: 0172 /2010
Record Dates: First submitted 2017-06-21; First posted 2017-11-21 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Late Onset Alzheimer Disease
Keywords: Alzheimer; APOE; CYP2D6; Donepezil; Genetics
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample was drawn from the patients on the first consultation for use in DNA extraction and Apolipoprotein E (APOE) genotyping. For the patients who were taking donepezil, after three, six and twelve months of treatment another blood sample were also drawn, separated in plasma and kept into the freezer at - 70 Celsius degree for further analysis of serum level of donepezil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pharmacological treatment of AD is currently based on cholinesterase inhibitors (ChEI) and memantine, which have been shown to lead to modest, although effective, clinical benefits. Donepezil is a ChEI metabolized through the cytochrome P (CYP) 450, primarily by the 3A4 and 2D6 isoforms. The CYP2D6 gene presents polymorphisms that can alter its expression. The plasma therapeutic level ranges from 30 to 75 ng/mL, and 50% of acetylcholinesterase inhibition is achieved when the concentration reaches 15.6 ng/mL. An optimal plasma level is greater than 50 ng/mL.

These polymorphisms may influence the individual's response to treatment with donepezil and the concentration of the drug in AD patients, without achieving the desired effect. However, most of the individuals are EM, i.e., the metabolism of the drug occurs according to the expected kinetics and is associated with the presence of one or two wild-type alleles.

Objective: investigate the pattern of clinical response to donepezil in a group of patients with AD and AD with cerebrovascular disease (CVD) in relation to the plasmatic concentration of donepezil and polymorphisms of the CYP2D6 and apolipoprotein E (APOE) genes.

DETAILED DESCRIPTION:
Patients taking donepezil were seen four times (from June 2009 to March 2013) and were submitted to the MMSE test, the Consortium to Establish a Registry for Alzheimer'sDisease battery (CERAD), and the Pfeffer Functional Activities Questionnaire. CERAD memory evaluation was further divided into five components: incidental recall (CERAD151 INC), immediate recall 1 and 2 (CERAD-RM1, CERAD-RM2, respectively) and delayed recall after five minutes (CERAD-R). Each aspect was analyzed individually and compared between groups at baseline and after 12 months of treatment with donepezil. All patients had blood samples (10mL) collected to obtain donepezil plasmatic concentration (DPC) measurements and for APOE and CYP2D6 genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the National Institute on Aging and the Alzheimer's Association diagnostic criteria of probable AD dementia or the NINDS-AIREN (National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherché et l'Enseignement en Neurosciences) diagnostic criteria of AD with cerebrovascular disease (AD + CVD)
* Patients presenting mild or moderate dementia according to the Clinical Dementia Rating (CDR), i.e., CDR 1 or 2, respectively

Exclusion Criteria:

* Patients treated with ChEI or memantine before study entry
* Patients diagnosed with frontotemporal dementia, dementia with Lewy bodies or vascular dementia,
* Patients classified as CDR 3 or with Mild Cognitive Impairment
* Illiterate patients
* Disagreement between the first investigator and the treating physician regarding the diagnosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A longitudinal, naturalist study, conducted at the Geriatric Outpatient Clinic of the Hospital das Clínicas at the Federal University of Minas Gerais (UFMG), in Belo Horizonte (MG), Brazil.
  The sample comprised patients evaluated from June, 2009 until March, 2013
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Association among donepezil serum concentration after 3, 6, and 12 months of treatment onset and clinical response. | September, 2009 until March, 2013
  Evaluate the serum concentration of donepezil after 3, 6, and 12 months of treatment onset in patients considered good responders (i.e., those who had an increment >1 in MMSE in comparison to baseline assessment after 1 year of donepezil treatment) in contrast to those considered bad responders (i.e., who had a reduction, a stabilization or an increment of 1 in MMSE in comparison to baseline assessment after 1 year of donepezil treatment).

SECONDARY OUTCOMES:
Evaluation of baseline cognitive performance | June, 2009 until March, 2012
  Assess the baseline cognitive performance among included patients (notedly, MMSE test, CERAD batteries, and in the Pfeffer Functional Activities Questionnaire).
Evaluation of CYP2D6 and APOE polymorphisms | June, 2009 until March, 2012
  Evaluation of CYP2D6 and APOE polymorphisms among included patients.
Evaluate donepezil serum concentration after 3 months of treatment onset. | September, 2009 until June, 2012
  Measurement of donepezil serum concentration after 3 months of treatment onset.
Evaluate donepezil serum concentration after 6 months of treatment onset. | December, 2009 until September, 2012
  Measurement of donepezil serum concentration after 6 months of treatment onset.
Evaluate donepezil serum concentration after 12 months of treatment onset. | June, 2010 until March, 2013
  Measurement of donepezil serum concentration after 12 months of treatment onset.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Caramelli, MD, PhD, Study Chair — Federal University of Minas Gerais